CLINICAL TRIAL: NCT06079112
Title: A Phase Ib/II, Open-label, Single Arm, Multicenter Clinical Study to Evaluate the Safety and Efficacy of 9MW2821 Combined With Toripalimab Injection in Subjects With Local Advanced or Metastatic Urothelial Cancer
Brief Title: 9MW2821 Combined With Toripalimab Injection in Subjects With Local Advanced or Metastatic Urothelial Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9MW2821-2023-CP104
Record Dates: First submitted 2023-09-25; First posted 2023-10-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-10

CONDITIONS: Advanced Urothelial Carcinoma
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 9MW2821+Toripalimab (Experimental)
  Interventions: Drug: 9MW2821; Drug: Toripalimab

INTERVENTIONS:
Drug: 9MW2821 — 1.0/1.25/1.5 mg/kg, intravenous (IV) infusion every cycle until disease progression or intolerable toxicity, etc.
  Other Names: 9MW2821 injection
Drug: Toripalimab — 240mg intravenous (IV) infusion every cycle until disease progression or intolerable toxicity, etc.
  Other Names: Toripalimab injection

SUMMARY:
This is a phase Ib/II, open-label, multicenter clinical study to evaluate the safety, tolerability, efficacy, pharmacokinetics and immunogenicity of 9MW2821 combined with Toripalimab injection in subjects with local advanced or metastatic urothelial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Sign and date the informed consent form e approved by independent ethics committe.
* Male or female subjects aged 18 to 80 years (including 18 and 80 years).
* ECOG status of 0 or 1.
* Histologically or cytologically confirmed local advanced or metastatic urothelial cancer
* Subjects have received at least 1 line advanced standard therapy or were not treated before
* Subjects must submit tumor tissues for test
* Life expectancy of ≥ 12 weeks.
* Subjects must have measurable lesions according to RECIST (version 1.1).
* Adequate organ functions
* Sexually active fertile subjects, and their partners, must agree to use methods of contraception during the study and at least 6 months after termination of study therapy.
* Subjects are willing to follow study procedures.

Exclusion Criteria:

* Anti-tumor treatment such as chemotherapy and radiotherapy within 21 days prior to the first dose of study drug.
* Major surgery within 28 days prior to first dose of study drug.
* PD-1/PD-L1/PD-L2 inhibitors used in the previous treatment for La/m UC.
* Previous treatment with ADCs conjugated with MMAE payload.
* Clinical significantly toxicity Grade ≥ 2 (except alopecia and pigmentation) related to previous treatment.
* Peripheral neuropathy Grade ≥ 2.
* Poorly controlled blood sugar.
* Increased risks of corneal disease assessed by the investigator prior to the first dose of study drug.
* Documented history of clinically significant cardiac or cerebrovascular diseases within 6 months prior to the first dose of study drug.
* Active infections, such as uncontrolled HBV/HCV/HIV/TB infection, etc.
* Other serious or uncontrolled diseases, such as serious interstitial pneumonia/asthma, serious thromboembolic events, etc.
* Poorly controlled central nervous system metastases.
* Organ transplantation or allogeneic hematopoietic stem cell transplantation in the past.
* History of drug abuse or mental illness.
* Known allergic sensitivity to any of the ingredients of the study drug.
* Any P-glycoprotein (P-gp) inducers/inhibitors or potent CYP3A4 inducers/inhibitors within 14 days prior to the first dose of study drug.
* History of autoimmune disease requiring systemic treatment within 2 years before the first dose.
* Any live vaccines within 4 weeks before first dose of study drug or during the study.
* Use of any investigational drug or medical instruments within 28 days prior to the first dose of study drug.
* History of another malignancy within 3 years before the first dose of study drug. Subjects with curable malignancies are allowed.
* Other conditions unsuitable into the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
incidence of AE/SAE | Up to 24 months
  adverse event(AE) 、serious adverse event(SAE)

SECONDARY OUTCOMES:
Objective Response Rate, ORR | Up to 24 months
  complete response (CR) or partial response (PR)
Duration of Response, DOR | Up to 24 months
  Time from the date of the first CR or PR to the earliest date of disease progression or death
Time To Response, TTR | Up to 24 months
  Time from the date of first infusion to the date of CR or PR
Disease Control Rate, DCR | Up to 24 months
  the percentage of subjects who experience CR, PR or stable disease (SD)
Progression-Free Survival, PFS | Up to 24 months
  Time from the date of first infusion to the earliest date of disease progression or death
Overall Survival, OS | Up to 24 months
  Time from the date of first infusion to the date of death
Pharmacokinetics parameter | Up to 12 months
  drug concentration of 9MW2821
Immunogenicity parameter | Up to 12 months
  Anti-Drug Antibody (ADA) of 9MW2821

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China